CLINICAL TRIAL: NCT05834036
Title: Effect of Antibiotics on Submucosal Enteric Neurons and Glia in the Lower Gastrointestinal
Brief Title: Effect of Antibiotics on Enteric Neurons and Glia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Yelina Alvarez, Principal Investigator, Rockefeller University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: YAL-1038
Record Dates: First submitted 2023-04-14; First posted 2023-04-28 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Antibiotic Enterocolitis
Keywords: Glia; Enteric Neurons
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Healthy Controls (Experimental): Healthy controls
  Interventions: Drug: Amoxicillin Oral Capsule

INTERVENTIONS:
Drug: Amoxicillin Oral Capsule — Amoxicillin 875mg every 12 hours for 7 days.
  Other Names: Amoxacillin oral capsule

SUMMARY:
The interactions between bacteria and their products with the intestinal tissue are important for maintaining a healthy and balanced system. Alterations in gut bacteria communities have been associated with various human pathologies. The investigators have found that mice treated with short and long-term antibiotics exhibit a transient yet profound loss of neurons in the more superficial submucosal and deeper muscularis plexi in the intestine accompanied by slow motility. Glia cells also depend on microbiota for their maintenance. In humans, antibiotic use has been associated with disorders of gut-brain interactions (DGBI) such as irritable bowel syndrome however whether there are changes in the enteric neurons and glia cells remain unknown. Therefore, the investigators propose to further characterize the neurons and glia populations in the human distal colon after a single antibiotic course. This study will reveal glia and neuronal subtypes that are susceptible to changes in the bacteria populations and depend on microbial products for their maintenance. These findings will guide future DGBI studies to ascertain the physiological effects that such loss has on intestinal healthy balance.

DETAILED DESCRIPTION:
The enteric nervous system (ENS) has been recognized as the "second brain" as it can regulate enteric physiology without central nervous system input. Similar to the central nervous system, it is composed of multiple neuron populations whose main functions are gut motility, secretion, and absorption. In addition to the neurons, the ENS contains glia cells whose main role is neuroprotection but also contribute to normal gut motility. Several studies have demonstrated that the microbiota and the ENS have an intimate relationship that begins in utero, and it is critical for its normal development. Neurons can recognize bacteria and their products. Several investigators have shown neuronal loss after enteric infections and antibiotic (Ampicillin) treatment in the muscularis layer, that results in delayed transit time in animal models. Hence, communication between the microbiota and the ENS is important to maintain normal gut motility. Disorders of Gut-Brain Interactions (DGBIs) are quite common, among these are Irritable Bowel Syndrome (IBS) defined by Rome IV criteria as abdominal pain associated with a change in consistency and frequency of bowel movements and the constipation predominant subtype (less than 3 bowel movements per week) is the most prevalent, which is also the most common motility disorder that mouse models of infection and antibiotics treatment exhibit. IBS has been associated with dysbiosis and a recent study demonstrated that antibiotic use immediately before or after screening colonoscopy increased the risk of developing IBS. In addition, dysfunction of submucosal neurons in IBS has been previously reported but whether there are changes in neuron numbers or neuron characteristics has not been explored. While there have been prospective studies that have explored the effects of antibiotics in patients treated for Helicobacter Pylori, there have been other investigators who have focused on the long term effects of antibiotics in healthy volunteers.

Therefore, similar to animal models, investigators propose that humans experience a profound and transient loss/alteration of neurons in the setting of antimicrobial use associated dysbiosis that manifest as DGBIs, most notably the constipation subtypes. This proposal will address whether antimicrobial use leads to quantitative and qualitative changes in the populations of submucosal neurons and glia cells in human subjects.

This hypothesis will be tested in a prospective study in which healthy participants will be asked to take the commonly used antibiotic amoxicillin twice a day for 7 days, and colon tissue biopsies will be obtained before and after treatment. Human tissue will be processed and analyzed to visualize structural changes, and changes in gene expression, bacteria, metabolites will be determined through single nuclei RNA sequencing, 16S ribosomal bacteria RNA sequencing and metabolomics analysis respectively.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old of different sex and races.

Exclusion Criteria:

* Allergy to penicillin, amoxicillin, augmentin, ampicillin, and other antibiotics in the penicillin family
* Pregnancy or fertility treatments
* Usage of antibiotics, antifungals or antivirals within three months prior to participation
* Change in dietary habits within the last three months prior to participation such as transitioning from high fat western diet to primarily plant based diet, initiation of ketogenic, paleo or any other weight loss regimen.
* Acute (in the past 30 days) or chronic enteric infections, including C. difficile.
* Chronic gastrointestinal disorder including inflammatory bowel disease, celiac disease , irritable bowel syndrome, chronic constipation or diarrhea
* Active neuropsychiatric disorder that requires anti-psychotic ie typical and atypical antipsychotics as well as anti-epileptics, levodopa, rivastigmine or any other neuropsychiatric medication with dopaminergic and cholinergic effects.
* Myocardial infarction or cerebrovascular accident in the six months prior to participation
* Coagulation disorders
* Chronic immunosuppressive medication (systemic) usage
* Anti-coagulation and anti-platelet agents such as plavix, warfarin, heparin, direct oral anticoagulants.
* Low dose Aspirin does not constitute an exclusion criteria.
* Prior episode of C. difficile infection.
* Prosthetic heart valves or any other conditions that require pre-procedure antibiotics.
* Currently receiving chemotherapy
* Any medical, psychological or social condition, in the opinion of the investigator, would jeopardize the health or well-being of the participant, interfere with their participation in the study, or confound the results of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Number of colonic submucosal neurons in the colon | 1 year
  Total number of colonic submucosal neurons counted per mm^2 before and after antibiotics treatment.
Number of colonic submucosal glia in the colon | 1 year
  Total number of colonic submucosal glia counted per mm^2 before and after antibiotics treatment.

SECONDARY OUTCOMES:
Changes in gene expression in submucosal neurons | 1 year
  Neurons nuclei will be isolated, and RNA will be sequenced and identified through alignment to human genome. The amount of RNA will be normalized as transcripts per million (TPM unit) and fold changes of a transcript will be calculated by dividing the TPM numbers of a transcript before and after antibiotics treatment.
Changes in gene expression in submucosal glia | 1 year
  Glia nuclei will be isolated, and RNA will be sequenced and identified through alignment to human genome. The amount of RNA will be normalized as transcripts per million (TPM unit) and fold changes of a transcript will be calculated by dividing the TPM numbers of a transcript before and after antibiotics treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yelina Alvarez, MD/PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No